CLINICAL TRIAL: NCT00754169
Title: Warfighter Head Injury Study a Comprehensive, Multidisciplinary Research Evaluation
Brief Title: Warfighter Head Injury Study
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: United States Department of Defense (U.S. Federal Agency); National Institutes of Health Clinical Center (CC) (NIH); Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080198; 08-N-0198
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-01-09

CONDITIONS: Head Injury
Keywords: Traumatic Brain Injury; Brain Imaging; Brain Plasticity; Neuroplasticity; Neuropsychological Testing; Head Injury; Healthy Volunteer
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will examine the long-term outcome of brain injuries, the effects of treatment on outcome and the effects of brain injury on people s behavior and abilities.

Men and women between 18 and 75 years of age who served in combat in the Iraq war may be eligible for this study. It will compare test results in those who sustained a traumatic penetrating or blast-related brain injury during combat with those who did not.

Participants undergo the following procedures over a 5-day period of testing that lasts about 6 hours a day:

* Medical history and physical examination.
* Blood test for genetic analysis.
* Electroencephalography (EEG) to measure the electrical activity of the brain.
* MRI or CT scans of the brain to look at the structure and blood flow of the brain.
* Functional near-infrared spectroscopy (fNIRS) to monitor blood flow in the front part of the brain blood by measuring changes in near-infrared light.
* Neuropsychological testing, including questionnaires, pen-and-paper or computerized tests, and performance of simple actions to measure brain function, language, memory and other cognitive abilities..

DETAILED DESCRIPTION:
The Warfighter Head Injury Study (WHIS) is a comprehensive, multidisciplinary research study of head-injured warfighters to be conducted at the National Institutes of Health (NIH) in Bethesda, Maryland. The goals of the WHIS include providing clinicians and scientists with new insights into the short term recovery of function following traumatic brain injury (TBI), the role of the prefrontal cortex (PFC) in executive and social functions, and to identify better predictors of short term outcome (including cognitive, neurological, and genetic factors). With the assistance of the Department of Veterans Affairs/Veterans Health Administration (VA/VHA), we propose to contact all Iraqi-Afghan (IA) warfighters with penetrating head injury (PHI), a cohort of blast injured warfighters, and a group of matched (for time in service, combat exposure, age, gender, and preinjury Armed Services Vocational Aptitude Battery [ASVAB] scores) healthy warfighter controls as well as healthy volunteers with different blast exposures (i.e.: explosives experts, artillery operators, etc ) but no documentation of brain injury. We will inquire about their willingness to participate in a comprehensive, multidisciplinary outpatient evaluation conducted at the NIH. In addition to IA warfighters, we also plan to enroll Vietnam warfighters who were included in the W. F. Caveness Vietnam Head Injury Study (VHIS) Registry, in order to conduct detailed comparisons between groups. These cohorts represent a unique opportunity for study; they were healthy and employed before injury, preinjury intelligence testing is available, and the VA/VHA permits long-term follow-up. We have previously investigated Vietnam warfighters with PHI and the published results of those studies have changed the management and evaluation of head-injured warfighters, and contributed to knowledge of brain function and the long-term effects of head injury. Furthermore, based on the knowledge acquired in our previous research with Vietnam warfighters and our current interests in the functions of the human PFC, cognitive neuroplasticity in the young brain, posttraumatic stress disorder (PTSD), posttraumatic epilepsy (PTE), caregiver stress, and genetic-plasticity relationships, we are proposing a series of new cognitive neuroscience experiments and battery of standardized neuropsychological testing to be conducted during the WHIS. In this effort, the experimental testing will be complemented with structural imaging (magnetic resonance imaging [MRI] or computed tomography [CT]), diffusion tensor and perfusion imaging, electroencephalogram (EEG), near-infrared spectroscopy (NIRS), and molecular genetics evaluations. This combination of unique patients, cutting edge cognitive neuroscience experiments and state of the art techniques will lead to new scientific knowledge and improved clinical management of warfighters with TBI.

ELIGIBILITY:
-

TBI PATIENTS:

We will study up to 320 head-injured IA warfighters (200 PHI and 120 blast injuries), most of whom have served in Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF), and up to 500 who have been included in the VHIS Registry. PHI makes up about 20% of the total TBI from OIF and OEF.

We will ask all WHIS patients to travel to the NIH with their primary caregiver to serve as their Durable Power of Attorney (DPA) (see Section X for more information on the DPA); Caregivers will be asked to complete questionnaires and will execute a separate consent (see Caregiver Consent Form).

Inclusion of active duty military personnel is not essential to this study and can be completed without them, if necessary.

INCLUSION:

* Both sexes will be included, however we expect the cohort to be overwhelmingly (>90%) male,
* Age range18-75;
* At least 6 months post-head injury; or
* Those patients who have previously participated in the VHIS.

EXCLUSION:

-Any medical condition that, in the judgment of investigators, would make participation detrimental to the patient (e.g.: severe clinical depression, unstable heart disease).

CONTROLS:

We will recruit 50 of the VHIS controls, 200 healthy IA warfighter control subjects, with no history of neurologic or serious psychiatric disorder or any other medical condition that would pose a risk from participation (e.g., unstable heart disease) and 120 healthy volunteers with different exposures but no documentation of brain injury. An example of this latter group would include someone who might be employed as a teacher of the proper use of explosive devices (i.e. a trainer from the Bureau of Alcohol, Tobacco and Firearms) and functions well in that position except for an occasional complaint. We will recruit up to a total of 370 normal volunteers.

We will ask all WHIS controls to travel to the NIH with a companion, some one deemed close to them in terms of relationship (i.e.spouse, child, etc.), to serve as control participants for the caregivers of warfighters. Companions will be asked to complete questionnaires and will execute a separate consent (see Caregiver/Companion Consent Form).

INCLUSION:

* Control subjects will be healthy IA warfighter volunteers who are matched to head-injured IA warfighters for time in service, combat exposure, age, gender and preinjury ASVAB scores. All IA warfighter control participants must provide copies of their ASVAB induction testing scores, if applicable; or
* Individuals who have had different blast exposures (e.g., explosives expert) but no documentation of brain injury; or
* Those warfighter controls who have previously participated in the VHIS.

EXCLUSION:

* Neurological or psychiatric conditions as mentioned above;
* History of drug abuse; or
* Unable to travel independently.

CAREGIVERS/COMPANIONS:

We will enroll caregivers and companions (i.e.: family members, domestic partners, etc.) of WHIS Warfighter participants in order to learn more about the potential burden and related issues experienced by this group.

INCLUSION:

* Provides care to a Warfighter or,
* Chosen by a control participant as a close companion; and
* Their Warfighter provides informed consent and agrees to participate in the WHIS project.

EXCLUSION:

* Inability to provide informed consent; or
* No working knowledge of the English language.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2008-09-05; Study Completion 2013-01-09

PRIMARY OUTCOMES:
The effects of focal lesions on neuroplastic changes in cognitive and social functions following combat-related traumatic brain injury

SECONDARY OUTCOMES:
Genetic influence on neuroplastic changes in cognitive and social functions following combat-related traumatic brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abell F, Krams M, Ashburner J, Passingham R, Friston K, Frackowiak R, Happe F, Frith C, Frith U. The neuroanatomy of autism: a voxel-based whole brain analysis of structural scans. Neuroreport. 1999 Jun 3;10(8):1647-51. doi: 10.1097/00001756-199906030-00005. PMID 10501551
- [Background] Adolphs R. The neurobiology of social cognition. Curr Opin Neurobiol. 2001 Apr;11(2):231-9. doi: 10.1016/s0959-4388(00)00202-6. PMID 11301245
- [Background] Adolphs R. Cognitive neuroscience of human social behaviour. Nat Rev Neurosci. 2003 Mar;4(3):165-78. doi: 10.1038/nrn1056. PMID 12612630